CLINICAL TRIAL: NCT07341386
Title: Prevention of Recurrence of Herpes Simplex in Patients With Autoimmune Rheumatic Diseases
Brief Title: Prevention of Recurrence of Herpes Simplex in Autoimmune Rheumatic Diseases
Acronym: PRoHerpARD
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 87204225.7.0000.0068
Record Dates: First submitted 2026-01-05; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-10

CONDITIONS: Autoimmune Rheumatic Diseases; Recurrent Herpes Simplex; Prevention
Keywords: Herpes Simplex Virus; Acyclovir; Autoimmune Rheumatic Diseases; Rheumatology; Pediatric Rheumatology; Antiviral Suppressive Therapy; Infectious Disease Prevention
MeSH Terms: conditions — Herpes Simplex | interventions — Acyclovir

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ACV (Active Comparator): Patients with autoimmune rheumatic diseases and a history of recurrent HS will receive oral acyclovir 400 mg twice a day for 12 months.
  ARD patients will be randomly assigned in a 1:1 ratio, with the use of an automated Web and telephone system, to one of two subgroups: ACV or Placebo.
  Interventions: Drug: Acyclovir (ACV)
- Placebo (Placebo Comparator): Patients with autoimmune rheumatic diseases and a history of recurrent HS will receive oral placebo twice a day for 12 months.
  ARD patients will be randomly assigned in a 1:1 ratio, with the use of an automated Web and telephone system, to one of two subgroups: ACV or Placebo.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Acyclovir (ACV) — Oral acyclovir 400 mg twice a day for 12 months. Acyclovir is a synthetic nucleoside analog with in vitro activity against HSV-1, HSV-2, VZV, and other herpesviruses.
  Arms: ACV
Other: Placebo — Matching oral placebo, administered twice a day for 12 months.
  Arms: Placebo

SUMMARY:
The goal of this randomized, double-blind, placebo-controlled clinical trial is to evaluate the effectiveness and safety of oral suppressive therapy with acyclovir in preventing herpes simplex virus (HSV) reactivation in patients with autoimmune rheumatic diseases (ARDs) who have a history of recurrent HS episodes.

The main questions this study aims to answer are:

Does continuous oral acyclovir reduce the frequency of HSV reactivation in ARD patients compared to placebo? What is the safety profile of prolonged acyclovir use in this population? What are the main risk factors (clinical and treatment-related) associated with HSV reactivation in immunosuppressed patients.

Participants will:

Be randomly assigned (1:1) to receive oral acyclovir (400 mg BID) or placebo for 12 months; Be followed for a total of 24 months, with regular clinical evaluations (every 3 months) and laboratory monitoring (every 3 months); Be assessed for HSV recurrence based on clinical symptoms, detection of HSV DNA by polymerase chain reaction (PCR) in mucocutaneous swabs in doubtful cases, and standardized reporting forms; Undergo disease activity assessments and adverse event monitoring at regular intervals.

The study includes adult and pediatric patients with confirmed diagnoses of one of the following ARDs: systemic lupus erythematosus (SLE), rheumatoid arthritis (RA), juvenile idiopathic arthritis (JIA), ankylosing spondylitis (AS), psoriatic arthritis (PsA), dermatomyositis/polymyositis (DM/PM), systemic sclerosis (SSc), systemic vasculitis, primary Sjögren's syndrome, Mixed connective tissue disease (MCTD), Chronic recurrent multifocal osteomyelitis (CRMO), Sarcoidosis and Behçet's Syndrome. All participants must have a documented history of recurrent HSV (oral and/or genital) before inclusion.

DETAILED DESCRIPTION:
HSV-1 and HSV-2 are ubiquitous human pathogens that can establish lifelong latency, with the potential for frequent reactivation. Immunocompromised individuals, including patients with ARDs, are particularly vulnerable to more severe and disseminated HSV infections, which may result in significant morbidity and even mortality. Despite this, the true incidence and burden of HSV reactivation in ARD patients under immunosuppression remain underexplored.

Previous studies in solid-organ transplant recipients and people living with HIV have demonstrated that prophylactic or suppressive antiviral therapy with acyclovir can significantly reduce HSV-related complications. However, no randomized controlled trials to date have evaluated the efficacy and safety of this approach in ARD patients under frequent immunosuppressive drug use and recurrent HSV in this group.

This trial will enroll 62 participants with ARDs and prior recurrent HSV infection, randomly assigned to receive oral acyclovir or placebo for 12 months, followed by continued monitoring for an additional year. Primary outcomes include the number of clinically confirmed HSV reactivations in acyclovir and placebo groups. Secondary outcomes include safety (adverse events), treatment tolerability, and identification of clinical and therapeutic risk factors for HSV recurrence.

By providing high-quality evidence through a rigorously controlled methodology, this study seeks to fill a critical knowledge gap in rheumatology, offering practical guidance for antiviral prophylaxis in immunosuppressed ARD patients, ultimately improving patient safety and clinical outcomes in a vulnerable population.

ELIGIBILITY:
Inclusion Criteria

* Eligible participants must be >12 years old, of any sex, and have a confirmed diagnosis of an autoimmune rheumatic disease (ARD) based on internationally accepted classification criteria, including rheumatoid arthritis (ACR/EULAR 2010), juvenile idiopathic arthritis (ILAR), axial spondyloarthritis (ASAS 2009), psoriatic arthritis (CASPAR 2012), systemic lupus erythematosus (SLICC 2012), systemic sclerosis (ACR 2013), dermatomyositis/polymyositis (Bohan & Peter), systemic vasculitis (Takayasu arteritis, granulomatosis with polyangiitis, polyarteritis nodosa), primary Sjögren's syndrome (ACR/EULAR 2016), mixed connective tissue disease (Alarcón-Segovia or Kasukawa criteria), chronic recurrent multifocal osteomyelitis (Jansson et al., 2007), sarcoidosis (ATS/ERS/WASOG 2020 statement), and Behçet's syndrome (International Study Group, 1990).
* Eligible patients must present serologic evidence of prior HSV infection (complement fixation titer ≥ 1:8) and a clinical history of recurrent oral or genital herpes simplex virus infection, defined as at least four episodes in the past 12 months.

Exclusion Criteria

- Participants will be excluded if they have a known hypersensitivity to acyclovir or any component of the study medication.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2026-01-05 (Estimated); Primary Completion 2027-12-01 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
HSV Reactivation Rate | Baseline to Month 24
  Proportion of patients with autoimmune rheumatic diseases (ARDs) and history of recurrent HS who experience clinical reactivation of HSV (oral and/or genital) during the 12-month treatment period and during the following 12 months. Reactivation will be defined by clinical signs and symptoms of HS, detection of HSV DNA by PCR in mucocutaneous swabs in doubtful cases.

SECONDARY OUTCOMES:
Safety Profile - Adverse Events (AEs) | Day 1 through Month 12
  Frequency and severity of adverse events (e.g., gastrointestinal discomfort, headache, rash) reported during the 12-month treatment phase.
Frequency of Serious Adverse Events (SAEs) | Day 1 through Month 12
  Incidence of SAEs (hospitalization, death, drug-related complications) in the acyclovir and placebo groups.
Treatment Discontinuation Due to AEs | Day 1 through Month 12
  Proportion of participants who discontinue acyclovir or placebo due to adverse events.
Time to First HSV Reactivation | Day 1 through Month 12
  Number of days from randomization to first documented HSV reactivation.
Factors Associated with HSV Reactivation | Day 1 through Month 24
  Analysis of clinical (disease activity) and treatment-related factors (e.g., corticosteroid dose, immunosuppressive drugs and biologic therapy) associated with increased risk of HSV reactivation.
Disease Activity Flares - Systemic Lupus Erythematosus | Day 1 through Month 12
  Systemic Lupus Erythematosus (SLE): An increase of more than three points in the Systemic Lupus Erythematosus Disease Activity Index 2000 (SLEDAI-2K).
Disease Activity Flares - Rheumatoid Arthritis | Day 1 through Month 12
  Rheumatoid Arthritis (RA): An absolute increase in Disease Activity Score - C-reactive protein (DAS28-CRP) > 1.2, or an increase in DAS28-CRP > 0.6 if baseline DAS28-CRP > 3.2.
Disease Activity Flares - Juvenile Idiopathic Arthritis | Day 1 through Month 12
  Juvenile Idiopathic Arthritis (JIA): An increase in Juvenile Arthritis Disease Activity Score (JADAS-27) > 5 points, or clinical worsening of ≥ 2 active joints requiring therapy escalation, in accordance with ACR Pediatric Response criteria.
Disease Activity Flares - Ankylosing Spondylitis | Day 1 through Month 12
  Ankylosing Spondylitis (AS): An increase in Ankylosing Spondylitis Disease Activity Score (ASDAS) > 0.9.
Disease Activity Flares - Psoriatic Arthritis | Day 1 through Month 12
  Psoriatic Arthritis (PsA): Worsening in disease activity classification by Disease Activity Index for Psoriatic Arthritis (DAPSA). If the patient was already in the worst status, clinical judgment and therapy increments were applied. For the following diseases, the definition of flare relied on clinical judgment and the need for increased therapy, supported by various disease scores.
Disease Activity Flares - Dermatomyositis/Polymyositis | Day 1 through Month 12
  Dermatomyositis/Polymyositis (DM/PM): Based on the International Myositis Assessment and Clinical Studies Group (IMACS) core set: Myositis Disease Activity Assessment (MYOACT), Health Assessment Questionnaire (HAQ), Patient's and Physician's Visual Analog Scales (VAS), ACR/EULAR Myositis Response Criteria (MRC) and the MMT8.
Disease Activity Flares - Systemic Sclerosis | Day 1 through Month 12
  Systemic Sclerosis (SSc): Increase in the modified Rodnan skin score, development of new digital ulcers, worsening dyspnea classified by NYHA functional scale, or increase in the EULAR Systemic Sclerosis Impact of Disease Index (ScleroID).
Disease Activity Flares - Systemic Vasculitis | Day 1 through Month 12
  Systemic Vasculitis (ANCA-associated vasculitis, including granulomatosis with polyangiitis, eosinophilic granulomatosis with polyangiitis, and microscopic polyangiitis): Increase in Birmingham Vasculitis Activity Score (BVAS).
Disease Activity Flares - Primary Sjögren's Syndrome | Day 1 through Month 12
  Primary Sjögren's Syndrome (SjD): EULAR Sjögren's Syndrome Disease Activity Index (ESSDAI).
Disease Activity Flares - Mixed Connective Tissue Disease | Day 1 through Month 12
  Mixed Connective Tissue Disease (MCTD): Increase in the Kahn & Appelboam MCTD Activity Score.
Disease Activity Flares - Chronic Recurrent Multifocal Osteomyelitis | Day 1 through Month 12
  Chronic Recurrent Multifocal Osteomyelitis (CRMO): Recurrence or emergence of ≥ 1 new bone lesion confirmed by MRI, or increase ≥ 2 points in the Pediatric/Adult CRMO Activity Score (PCAS/ACAS), accompanied by the need for escalation of anti-inflammatory or disease-modifying therapy.
Disease Activity Flares - Sarcoidosis | Day 1 through Month 12
  Sarcoidosis: Increase ≥ 2 points in the Sarcoidosis Activity Assessment Tool (SAAT) or worsening in the Sarcoidosis Clinical Activity Classification (SCAC), defined by recurrence or progression of pulmonary infiltrates, increase in serum ACE levels > 30%, or new extrapulmonary organ involvement requiring treatment intensification.
Disease Activity Flares - Behçet's Syndrome | Day 1 through Month 12
  Behçet's Syndrome: Based on the Behçet's Disease Current Activity Form simplified version (BDCAF-s), considering recurrence of oral or genital ulcers, new ocular inflammation, vascular or neurological involvement, or any increase ≥ 2 points in BDCAF-s global score.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ioannidis JP, Collier AC, Cooper DA, Corey L, Fiddian AP, Gazzard BG, Griffiths PD, Contopoulos-Ioannidis DG, Lau J, Pavia AT, Saag MS, Spruance SL, Youle MS. Clinical efficacy of high-dose acyclovir in patients with human immunodeficiency virus infection: a meta-analysis of randomized individual patient data. J Infect Dis. 1998 Aug;178(2):349-59. doi: 10.1086/515621. PMID 9697714
- [Background] Fatahzadeh M, Schwartz RA. Human herpes simplex virus infections: epidemiology, pathogenesis, symptomatology, diagnosis, and management. J Am Acad Dermatol. 2007 Nov;57(5):737-63; quiz 764-6. doi: 10.1016/j.jaad.2007.06.027. PMID 17939933
- [Background] Beyar-Katz O, Bitterman R, Zuckerman T, Ofran Y, Yahav D, Paul M. Anti-herpesvirus prophylaxis, pre-emptive treatment or no treatment in adults undergoing allogeneic transplant for haematological disease: systematic review and meta-analysis. Clin Microbiol Infect. 2020 Feb;26(2):189-198. doi: 10.1016/j.cmi.2019.09.003. Epub 2019 Sep 16. PMID 31536817